CLINICAL TRIAL: NCT05828849
Title: Can a Radical Transformation of Preventive Care Reduce Mortality by 20% in Low Socioeconomic (SES) Populations? Preparatory Work Focusing on Alcohol Use Disorder (AUD)/Heavy Alcohol Use, HIV Risk, and Cardiovascular Risk
Brief Title: Mortality Reductions Based on AUD/Heavy Alcohol Use, HIV Risk, and Cardiovascular Risk
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-01584
Record Dates: First submitted 2023-04-13; First posted 2023-04-25 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-04

CONDITIONS: Cardiovascular Disease; Alcohol Use Disorder; HIV Risk; Substance Use Disorders
MeSH Terms: conditions — Cardiovascular Diseases; Alcoholism; Substance-Related Disorders | interventions — Compensation and Redress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low SES Population - Intervention (Experimental): Participants receive the study intervention, composed of navigation, compensation, and personalization for study participants. The intervention will be administered in person to the participants recruited for the study and will be administered by peer navigators who will be trained on Motivational Interviewing (MINT) techniques.
  Interventions: Behavioral: Navigation, compensation, and personalization
- Low SES Population - No Intervention (No Intervention): Participants receive no intervention components of navigation, compensation, and personalization. Participants will receive their normal medical care through regular doctor visits without any intervention or personalization.

INTERVENTIONS:
Behavioral: Navigation, compensation, and personalization — The study intervention is composed of navigation, compensation, and personalization. Navigation refers to reducing barriers posed by fragmentation of health and social systems. Compensation refers to reimbursement of out-of-pocket expenses to offset dependent care, time costs, and travel expenditures necessary to access care for the different conditions and goals of the intervention. Personalization refers to preventative interventions that are personalized based on individual for potential benefit.
  Arms: Low SES Population - Intervention

SUMMARY:
The purpose of this research study is to investigate if a personalized intervention including parts such as navigation (focus on patient outreach efforts, missed and completed encounters), personalization (individual health benefits) and compensation (value health-related costs borne by patients) will help people reduce their chances of dying from preventable causes, including heart attacks, strokes, drinking alcohol, substance abuse, HIV, and other conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Age 35 to 64
2. Low SES (≤ $38,000 annual income, based on 2019 20th percentile NYC income, adjusted for family size)
3. Expected mortality ≥1% per year (based on age, sex, race/ethnicity), with ≥1 of the following contributors:

   1. 10-year cardiovascular risk ≥10% (assessed by ASCVD risk tool)
   2. Heavy alcohol consumption (defined using SAMHSA binge drinking definition, drinking >4 standard drinks for men and >3 standard drinks for women on same occasion in past month)
4. Willing to be navigated to Health and Hospitals Corporation of New York health system.
5. Ability to provide written informed consent in English or Spanish

Exclusion Criteria:

1. Receives regular care elsewhere than Health and Hospitals Corporation of New York
2. Already diagnosed with high mortality-condition(s) that are not included in the simulation model.

Ages: 35 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2024-06-25 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in Alcohol Use Disorders Identification Test (AUDIT) Score | Baseline, Month 12
  10-item self-assessment of alcohol use disorders. Items are rated on a scale from 0 to 4. The total score is the sum of responses and ranges from 0-40; higher scores indicate it is more likely the patient's drinking is affecting their health and safety.
Change in Alcohol Use Disorders Identification Test-Concise (AUDIT-C) | Baseline, Month 12
  4-item self-assessment of alcohol use disorders. Items are rated on a scale from 0 to 4. The total score is the sum of responses and ranges from 0-12; higher scores indicate it is more likely the patient's drinking is affecting their health and safety.
Change in National Institute on Alcohol Abuse and Alcoholism (NIAAA) single-item alcohol use screen (NIAAA-1) | Baseline, Month 12
  The NIAAA-1 asks participants how many times in the past year they have had four or more drinks (for females) or five or more drinks (for males) in a day. The responses are 0 (never), 1 (Less than once a month), 2 (One to three times per month), 3 (One to three times per week) and 4 (More than three times per week). The total score is the item response and ranges from 0-4; higher scores indicate greater unhealthy alcohol use.
Change in 2-Week Timeline Follow-Back (TLFB) for Alcohol Use | Baseline, Month 12
  The TLFB allows participants to indicate how many drinks they have had over the previous two weeks.
Change in Ethanol Glucuronide (ETG) Levels | Baseline, Month 12
  ETG (ng/ml) will be measured via urine test.
Change in Phosphatidylethanol (PeTH) Levels | Baseline, Month 12
  PeTH (ng/ml) will be measured via blood test.
Change in CDC HIV Incidence Risk Index Score | Baseline, Month 12
  3-item assessment of HIV risk among people who inject drugs. The total score ranges from 0 to 100; higher scores indicate greater risk of HIV.
Change in American Heart Association/American College of Cardiology (AHA/ACC) ASCVD Risk Calculator Score | Baseline, Month 12
  The AHA/ACC Atherosclerotic Cardiovascular Disease (ASCVD) Risk Calculator is a questionnaire that uses responses to calculate the lifetime risk of ASCVD as a percentage (0%-100%); higher percentages indicate greater lifetime risk of ASCVD. The percentages are classified as follows:
  * Low-risk (<5%)
  * Borderline risk (5% to 7.4%)
  * Intermediate risk (7.5% to 19.9%)
  * High risk (≥20%)
Mean Systolic Blood Pressure | Up to Month 12
Mean Diastolic Blood Pressure | Up to Month 12
Percent Change in Participants Determined to be "High-Risk" for SUD per TAPS Screening Tool | Baseline, Month 12
  The Tobacco, Alcohol, Prescription medication, and other Substance use (TAPS) Tool is used to assess primary care patients for tobacco, alcohol, prescription drug, and illicit substance use and problems related to their use. Based on patient responses, the tool classifies the patient risk levels as "High Risk," "Problem Use," "Undetermined Risk" and "Minimal Risk." This outcome measures the percent change in participants determined to be "High Risk" for substance abuse disorder (SUD) from baseline to Month 12.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald S Braithwaite, Braithwaite, Principal Investigator — NYU Langone Health
Locations (1):
- NYC H+H/Bellevue, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: [Dr. Ronald Scott Braithwaite, Scott.Braithwaite@nyulangone.org]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Scott.Braithwaite@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

DOCUMENTS (1):
  • Informed Consent Form (2023-03-29): https://cdn.clinicaltrials.gov/large-docs/49/NCT05828849/ICF_000.pdf